CLINICAL TRIAL: NCT04180371
Title: Phase I/II Study of the Safety, Pharmacokinetics, and Preliminary Clinical Activity of BT5528 in Patients With Advanced Malignancies Associated With EphA2 Expression
Brief Title: Study BT5528-100 in Patients With Advanced Solid Tumors Associated With EphA2 Expression
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BicycleTx Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT5528-100
Record Dates: First submitted 2019-11-19; First posted 2019-11-27 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor Historically Known for High EphA2 Expression; Urothelial Cancer; Ovarian Cancer; Non-small Cell Lung Cancer; Head and Neck Cancer; Triple Negative Breast Cancer; Gastric/Upper Gastrointestinal Cancer
Keywords: EphA2; ovarian cancer; urothelial cancer; bladder cancer; NSCLC; TNBC; gastric cancer; GEJ cancer; HNSCC
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Triple Negative Breast Neoplasms; Gastrointestinal Neoplasms; Urinary Bladder Neoplasms; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I - Dose escalation (BT5528) (Experimental): Cohorts of participants will receive increasing doses of BT5528. It is expected that up to 72 participants will participate in this dose escalation arm.
  Interventions: Drug: BT5528
- Phase I - Dose escalation combination (BT5528 & nivolumab) (Experimental): Cohorts of participants will receive increasing doses of BT5528 and a standard dose of nivolumab. It is expected that up to 24 participants will participate in this dose-escalation combination arm.
  Interventions: Drug: BT5528; Drug: Nivolumab
- Phase II - Dose expansion 1 (BT5528) (Experimental): A cohort of participants will receive the selected dose of BT5528 as a monotherapy. It is expected that up to 164 patients have solid tumors (Cohort 1: urothelial cancers, Cohort 2: ovarian cancer, Cohort 3: non-small cell lung cancer, Cohort 4: head and neck cancer, Cohort 5: triple-negative breast cancer, and Cohort 6: gastric/upper gastrointestinal cancer) historically known for high expression of EphA2 will participate in this dose-expansion arm, Cohort 7: urothelial MMAE exposed, Cohort 8: head and neck squamous cell carcinoma
  Interventions: Drug: BT5528

INTERVENTIONS:
Drug: BT5528 — Participants will receive a 60-minute intravenous infusion of BT5528 once a week (Days 1, 8, 15, and 22) or every other week (Days 1 and 15) on a 4-week cycle at the selected dose.
Drug: Nivolumab — Participants will receive nivolumab at 480mg intravenous infusion every 4 weeks.
  Other Names: Opdivo
  Arms: Phase I - Dose escalation combination (BT5528 & nivolumab)

SUMMARY:
This clinical trial is evaluating a drug called BT5528 alone and in combination with nivolumab in participants with advanced solid tumors historically known for expression of EphA2. The main goals of this study are to:

* Find the recommended dose(s) of BT5528 that can be given safely to participants alone and in combination with nivolumab
* Learn more about the side effects of BT5528
* Learn about how effective BT5528 is for the treatment of ovarian cancer, urothelial/bladder cancer, lung cancer (NSCLC), triple-negative breast cancer, head and neck cancer (HNSCC), and gastric/upper gastrointestinal cancer.
* Learn more about BT5528 therapy alone and in combination with nivolumab.

DETAILED DESCRIPTION:
BT5528 consists of a bicyclic peptide (Bicycle®) which binds to EphA2, and is covalently attached to a spacer and a protease cleavable peptide linker attached to MMAE.

The Phase I/II multi-center, open-label trial will evaluate BT5528 administered once-weekly as a single agent and in combination with nivolumab. The Phase I portion is a dose escalation primarily designed to assess the safety and tolerability of BT5528 and to determine recommended Phase II dose(s) (RP2D). Following selection of a recommended Phase II dose(s) (RP2D), a dose expansion portion will be initiated with the primary objective of evaluating the clinical activity of BT5528.

ELIGIBILITY:
General Inclusion:

* Written informed consent, according to local guidelines, signed and dated by the patient or by a legal guardian prior to the performance of any study-specific procedures, sampling or analyses
* At least 18 years-of-age at the time of signature of the informed consent form
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Acceptable renal, hepatic, hematologic and coagulation functions
* Negative pregnancy test for women of childbearing potential
* Male participants with female partners of childbearing potential and female participants of childbearing potential are required to follow highly effective contraception
* All patients must have tumor tissue (fresh or archived) available for analysis of EphA2 tumor expression and other biomarkers. In the absence of available tumor tissue, patients must be willing to undergo a biopsy to provide fresh tumor samples
* Life expectancy ≥12 weeks after the start of BT5528 treatment according to the Investigator's judgment.
* Must be willing and able to comply with the protocol and study procedures.

Additional inclusion criteria for Phase I (dose escalation phase, with BT5528 alone or in combination with nivolumab):

* Metastatic recurrent histologically confirmed malignant solid tumors historically known for high EphA2 tumor expression. Confirmation of EphA2 expression prior to enrollment is not required for participants with ovarian cancer and specific other individual tumor types.
* Exhausted all appropriate treatment options per local guidelines
* Participants with urothelial cancer who have at least 1 (but no more than 3) prior lines of systemic therapy.

Additional inclusion criteria for Phase II (dose expansion phase, with BT5528 alone):

* Participants with metastatic recurrent disease histologically confirmed to be non-small cell lung cancer, ovarian cancer, triple-negative breast cancer (TNBC), gastric/upper gastrointestinal (GI) cancer, head and neck (H&N) cancer, urothelial cancer are eligible and must have failed or are ineligible for all appropriate treatment options per local guidelines and must have evidence of radiographic progression on the most recent line of therapy
* Patients with urothelial cancer who have previously received treatment with enfortumab vedotin (EV) are eligible to the study. Patients who received EV and showed disease progression within 6 months of treatment start are planned for less than 50% of total patients enrolled in the cohort

Exclusion criteria (all participants):

* Chemotherapy treatments within 14 days prior to first dose of study treatment, other anticancer treatments, treatment within 28 days or 5 half-lives, whichever is the shorter
* Experimental treatments within 4 weeks of first dose of BT5528
* Prior toxicities must have resolved to Grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 (except alopecia which can be Grade 2), or well-controlled Grade 2 hypothyroidism or Grade 2 adrenal insufficiency on appropriate therapy
* Current treatment with strong inhibitors or inducers of CYP3A4 or strong inhibitors of P-gp
* Known sensitivity to any of the ingredients of the investigational product or monomethyl auristatin E (MMAE)
* Any condition, therapy or laboratory abnormality that might confound the results of the study, interfere with the patient's participation, or is not in the best interest of the patient to participate in the opinion of the investigator including but not limited to specific cardiovascular criteria
* Major surgery (excluding placement of vascular access) within 4 weeks of first dose of BT5528 study treatment and must have recovered adequately prior to starting study therapy
* Receipt of live vaccine within 30 days of study treatment
* Untreated CNS metastases or leptomeningeal disease
* Uncontrolled hypertension (systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg that is not responsive to intervention) at screening or prior to initiation of study drug.
* History or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the study, interfere with the patient's participation, or is not in the best interest of the patient to participate in the opinion of the Investigator including but not limited to:

  (a) Patients with history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, congestive heart failure or symptoms of New York Heart Association Class III-IV documented within 6 months prior to first dose of BT5528 or: (i) Mean resting corrected QT interval (QTcF) >470 msec (ii) Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval (iii) Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting electrocardiograms (ECGs), e.g., complete left bundle branch block, third degree heart block
* Known human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS). Note: Well controlled HIV will be allowed if the patient meets all the following criteria at inclusion:

  1. CD4+ T-cell (CD4+) counts ≥350 cells/uL;
  2. HIV viral load <400 copies/mL
  3. Without a history of opportunistic infection within the last 12 months.
  4. On established antiretroviral therapy (ART) for at least 4 weeks. Use of anti-retroviral therapy is permitted, but should be discussed with the Medical Monitor on a case-by-case basis.
* Patients with a positive hepatitis B surface antigen and/or anti-hepatitis B core antibody. Patients with a negative polymerase chain reaction (PCR) assay are permitted with appropriate antiviral therapy
* Active hepatitis C infection with positive viral load if hepatitis C virus (HCV) antibody positive (if antibody is negative then viral load not applicable). Patients who have been treated for hepatitis C infection can be included if they have documented sustained virologic response of ≥12 weeks.
* Thromboembolic events and/or bleeding disorders 3 months (e.g., deep vein thrombosis [DVT] or pulmonary embolism [PE]) prior to first dose
* Prior history of pneumonitis with presence of residual symptoms
* History of another malignancy within 3 years before the first dose of BT5528, or any evidence of residual disease from a previously diagnosed malignancy (excluding adequately treated with curative intent basal cell carcinoma, squamous cell of the skin, cervical intraepithelial neoplasia/cervical carcinoma in situ or melanoma in situ or ductal carcinoma in situ of the breast).
* Systemic anti-infective treatment or fever within the last 14 days prior to first dose of BT5528 study treatment
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.

Additional Exclusion Criteria (BT5528 in combination with nivolumab):

* Prior intolerance to immune checkpoint inhibitor
* Known hypersensitivity to checkpoint inhibitor therapy
* Prior organ transplant (including allogeneic)
* Diagnosis of clinically relevant immunodeficiency
* Active systemic infection requiring therapy
* More than 10 mg daily prednisone equivalent or other strong immunosuppressant
* History of autoimmune disease except alopecia, vitiligo, hypothyroidism, or adrenal insufficiency
* History of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Part A-1 and A-2(escalations): Number of participants receiving BT5528 alone and in combination with nivolumab with treatment-emergent adverse events | From Cycle 1 Day 1 (each cycle is 28 days) until 30 days post last dose
  Safety reported as incidence of treatment-emergent adverse events
Part A-1 and A-2 (escalations): Maximum tolerated dose (MTD) by the number of participants with dose limiting toxicities from BT5528 treatment alone and in combination with nivolumab | At the end of Cycle 1 (each cycle is 28 days)
  Maximum Tolerated Dose (MTD)
Part B: Objective response rate by RECIST 1.1 in participants with solid tumors historically known for high expression of EphA2 tumor expression receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks during study treatment)
  Objective Response Rate (ORR)
Part B: Duration of response by RECIST 1.1 in participants with solid tumors historically known for high expression of EphA2 receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks during study treatment)
  Duration of Response (DOR)
Part B: Clinical benefit rate by RECIST 1.1 in participants with solid tumors historically known for high expression of EphA2 receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks during study treatment)
  Clinical benefit rate
Part B: Time to tumor progression by RECIST 1.1 in participants solid tumors historically known for high expression of EphA2 receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks during study treatment)
  Time to Progression (TTP)
Part B: Progression-free survival by RECIST 1.1 in participants solid tumors historically known for high expression of EphA2 receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks during study treatment)
  Progression free survival (PFS)
Part B: PFS at 6 months by RECIST 1.1 in participants with solid tumors historically known for high expression of EphA2 receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months)
  Progression free survival (PFS)
Part B: Overall survival (OS) at 1 year in participants solid tumors historically known for high expression of EphA2 receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until death or loss of follow-up or withdrawal of consent
  Overall survival (OS)

SECONDARY OUTCOMES:
Part A-1 and A-2 (escalations): Objective response rate (ORR) by RECIST 1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 alone and in combination with nivolumab | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  Objective Response Rate (ORR)
Part A-1 and A-2 (escalations): Duration of response (DOR) by RECIST 1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 alone and in combination with nivolumab | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  Duration of Response (DOR)
Part A-1 and A-2 (escalations): Clinical benefit rate (CBR) by RECIST 1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 alone and in combination with nivolumab | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  Clinical benefit rate (CBR)
Part A-1 and A-2 (escalations): Time to tumor progression (TTP) by RECIST 1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 alone and in combination with nivolumab | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  Time to progression (TTP)
Part A-1 and A-2 (escalations): Progression-free survival (PFS) time by RECIST 1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 alone and in combination with nivolumab | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  Progression free survival (PFS)
Part A-1 and A-2 (escalations): Progression free survival at 6 months by RECIST 1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 alone and in combination with nivolumab | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months)
  Progression free survival (PFS)
Part A-1 and A-2 (escalations): Overall survival time at 12 months in participants with advanced solid tumors with high EphA2 levels receiving BT5528 alone and in combination with nivolumab | From Cycle 1 Day 1 (each cycle is 28 days) until death or loss of follow-up or withdrawal of consent (assessed every 3 months up to 12 months
  Overall survival (OS)
Part B: Determination of the number of participants with advanced solid tumors historically known for high expression of EphA2 receiving BT5528 with treatment-emergent adverse events | From Cycle 1 Day 1 (each cycle is 28 days) until 30 days post last dose
  Safety reported as incidence of treatment-emergent adverse events
All parts: Determine the plasma concentrations of BT5528 in plasma from all participants taking BT5528 alone and in combination with nivolumab | From Cycle 1,and end of each cycle (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or withdrawal of consent(assessed up to 12 months
  plasma concentrations of BT5528 in plasma from all participants taking BT5528 alone and in combination with nivolumab
All parts: Determine the plasma concentrations of MMAE in plasma from all participants taking BT5528 alone and in combination with nivolumab | From Cycle 1,and end of each cycle (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or withdrawal of consent(assessed up to 12 months
  plasma concentrations of MMAE in plasma from all participants taking BT5528 alone and in combination with nivolumab
All parts: Number of participants positive for anti-drug antibodies (ADA) from all participants receiving BT5528 alone and in combination with nivolumab | From Cycle 1,and end of each cycle (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or withdrawal of consent(assessed up to 12 months
Part B: The association between EphA2 expression level and objective response rate (ORR) per RECIST v1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  To investigate if the high expression of EphA2 is associated with high ORR per RECIST 1.1 participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment
Part B: The association between EphA2 expression level and duration of response (DOR) by RECIST 1.1 and per EphA2 expression in participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  To investigate if the high expression of EphA2 is associated with high DOR per RECIST 1.1 participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment
Part B: The association between EphA2 expression level and clinical benefit rate (CBR) per RECIST v1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  To investigate if the high expression of EphA2 is associated with high CBR per RECIST 1.1 participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment
Part B: The association between EphA2 expression level and time to tumor progression (TTP) per RECIST v1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  To investigate if the high expression of EphA2 is associated with long TTP per RECIST 1.1 participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment
Part B: The association between EphA2 expression level and progression-free survival (PFS) at 6 months by RECIST 1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until disease progression or death or new anti-cancer therapy or loss of follow-up or withdrawal of consent (assessed every 8 weeks up to 6 months then every 16 weeks up to 12 months
  To investigate if the high expression of EphA2 is associated with long PFS at 6 months per RECIST 1.1 participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment
Part B: The association between EphA2 expression level and overall survival (OS) at 1 year by RECIST v1.1 in participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment | From Cycle 1 Day 1 (each cycle is 28 days) until death or loss of follow-up or withdrawal of consent (assessed every 3 months up to 12 months)
  To investigate if the high expression of EphA2 is associated with long OS at 1 year per RECIST 1.1 participants with advanced solid tumors with high EphA2 levels receiving BT5528 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Meredith McKean, MD, MPH, Study Chair — Sarah Cannon and HCA Research Institute
Locations (28):
- United States (12):
  - California Cancer Associates for Research and Excellence, Inc., Encinitas, California
  - University of California - Irvine Medical Center, Orange, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Stephenson Cancer Center (Oklahoma University), Oklahoma City, Oklahoma
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital (UZA), Edegem
  - Universitair Ziekenhuis Gent (UZ), Ghent
- South Korea (2):
  - Gachon University Gil Medical Center, Incheon
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (5):
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
- United Kingdom (5):
  - Sarah Cannon Research Institute UK, London, United Kingdom
  - The Christie NHS Foundation Trust, Manchester, United Kingdom
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Leeds Teaching Hospitals NHS Trust Of Trust Headquarters, St James's University Hospital, Leeds
  - Sir Bobby Robson Cancer Trials Research Centre, The Northern Center for Cancer Care, Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No